CLINICAL TRIAL: NCT03464708
Title: A Study to Investigate the Effect of Eta-hydroxy-beta-methylbutyrate (HMB) on Skeletal Muscle Wasting in Early Critical Illness
Brief Title: A Study to Investigate the Effect of HMB on Skeletal Muscle Wasting in Early Critical Illness
Acronym: HMB-ICU
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17/LO/1635; 2016-003557-15 (EudraCT Number)
Record Dates: First submitted 2018-02-22; First posted 2018-03-14 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Critical Illness
Keywords: Critical illness; HMB; Nutrition; Muscle wasting; Recovery
MeSH Terms: conditions — Critical Illness; Muscular Atrophy | interventions — beta-hydroxyisovaleric acid; Lactose

STUDY DESIGN:
Intervention Model Description: Double blind, placebo controlled, randomised controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMB (Experimental): HMB 3 g/day until hospital discharge or 28-days (whichever comes first). HMB to be provided in powder form and administered via enteral feeding tube whilst in the ICU and orally once able to eat and drink.
  Interventions: Dietary Supplement: HMB
- Placebo (Placebo Comparator): Placebo (lactose) 3 g/day until hospital discharge or 28-days (whichever comes first). Placebo to be provided in powder form and administered via enteral feeding tube whilst in the ICU and orally once able to eat and drink.
  Interventions: Other: Lactose (placebo)

INTERVENTIONS:
Dietary Supplement: HMB — Powder form
  Other Names: beta-hydroxy-beta-methylbutyrate
  Arms: HMB
Other: Lactose (placebo) — Powder form
  Arms: Placebo

SUMMARY:
This study aims to investigate the effect of beta-hydroxy-beta-methylbutyrate (HMB) on skeletal muscle wasting, physical function, strength and quality of life in survivors of critical illness. In addition, protein turnover, muscle biology and muscle histology will be investigated.

DETAILED DESCRIPTION:
This is a double blind, placebo controlled, randomised controlled trial with the primary objective of investigating the effect of HMB on skeletal muscle wasting in early critical illness. Secondary objectives include determining the effect of HMB on skeletal muscle quality, strength, function and quality of life in survivors of critical illness. In addition, the effect of HMB on muscle protein turnover, muscle protein signalling, muscle fibre size and protein:DNA ratio will be investigated in a sub-group of participants.

Eligible participants will be randomised to receive either 3 g/day HMB or 3 g/day placebo within 24 hours of admission to the Intensive Care Unit (ICU). This will be continued until hospital discharge or 28-days, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

(i) ≥18 years old (ii) Due to receive enteral nutrition via a nasogastric or naso-jejunal tube as part of routine care (iii) Receiving mechanical ventilation and likely to continue this for more than 48 hours (iv) Likely to remain on the ICU for >7 days (v) Likely to survive intensive care admission. (vi) Admitted to recruiting ICU <24 hours from hospital admission and referring ICU ≥7 days from hospital admission (vii) Agreement obtained from legal representative (viii) Able to comply with protocol and study procedures (ix) No known allergy to IMP or any of its excipients

Participants in other trials can be recruited where protocols are not deemed likely to interfere with endpoints of either study and agreement has been obtained from the respective Chief Investigators.

Since participants in the trial will be abstaining by virtue of their illness, contraception is not required as an eligibility requirement.

Exclusion Criteria:

(i) Pregnancy or breast feeding (ii) Active disseminated malignancy (diagnosed) (iii) Bilateral lower limb amputees (iv) Non-ambulant or acute unilateral lower limb amputees (v) Patients with a primary neuromyopathy (vi) Patients entered into trials of interventions which would affect muscle mass (vii) Patients assessed as requiring sole parenteral nutrition (viii) Admission to ICU within the previous 3 months (ix) Any reason excluding ultrasound measurement being performed (x) Insufficient understanding of the trial by the legal representative (xi) Intolerance to lactose and/or milk protein allergy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change in rectus femoris cross-sectional area | Study Day 10
  Rectus femoris cross-sectional area will be measured using muscle ultrasound within 24 hours of admission to ICU and then again at study day 10. The difference between these measurements will then be determined.

SECONDARY OUTCOMES:
Change in rectus femoris cross-sectional area | Study day 7, ICU discharge (expected to be less than 10 days), hospital discharge or 28 days (whichever comes first), 3-months post-hospital discharge
  Rectus femoris cross-sectional area will be measured using muscle ultrasound within 24 hours of admission to ICU and then again at study day 7, ICU discharge, hospital discharge and 3-months post-hospital discharge. The difference between these measurements will then be determined.
Difference in muscle quality | Study day 7, study day 10, ICU discharge (expected to be less than 10 days), hospital discharge or 28 days (whichever comes first), 3-months post-hospital discharge
  Muscle quality will be measured determined by the echogenicity of the muscle, as measured using muscle ultrasound within 24 hours of admission to ICU and then again at study day 7,study day 10, ICU discharge, hospital discharge and 3-months post-hospital discharge. The difference between these measurements will then be determined.
Muscle strength | Study day 7, study day 10, ICU discharge (expected to be less than 10 days) and hospital discharge or 28 days (whichever comes first)
  Muscle strength will be measured using the Medical Research Council (MRC) Sum Score at study day 7, study day 10, ICU discharge and hospital discharge
Muscle strength | Study day 7, study day 10, ICU discharge (expected to be less than 10 days), hospital discharge or 28 days (whichever comes first), 3-months post-hospital discharge
  Muscle strength will be measured using handgrip dynamometry at study day 7, study day 10, ICU discharge, hospital discharge and 3-months post-hospital discharge
Physical function | Study day 7, study day 10, ICU discharge (expected to be less than 10 days), hospital discharge or 28 days (whichever comes first), 3-months post-hospital discharge
  Physical function will be measured using the Chelsea Physical Assessment Score (CPAx) at study day 7, study day 10, ICU discharge and hospital discharge.
Physical function | Hospital discharge or 28 days (whichever comes first), 3-months post-hospital discharge
  Physical function will be measured using the six-minute walk test at hospital discharge and 3-months post-hospital discharge.
Physical function | Hospital discharge or 28 days (whichever comes first), 3-months post-hospital discharge
  Physical function will be measured using the short physical performance battery (SPPB) at hospital discharge and 3-months post-hospital discharge.
Quality of life | 3-months post-hospital discharge
  Quality of life will be determined using the SF-36 survey at 3-months post-hospital discharge.
Inflammation, cell damage and metabolic profile | Study day 1, study day 7, study day 10
  Markers of inflammation, cell damage, and plasma metabolomics will be determined from plasma samples taken at study days 1, 7 and 10.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hart, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No